CLINICAL TRIAL: NCT06886828
Title: Virtual Reality Application During High Flow Nasal Oxygen Therapy in Children Effect on Anxiety Levels: A Randomised Controlled Study
Brief Title: Virtual Reality Application During High Flow Nasal Oxygen Therapy in Children Effect on Anxiety Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Tuğba Karakaya, Principal Investigator, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UskudarU-SBE-TK-01
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Distress
Keywords: high flow nasal oxygen therapy; virtual reality; Anxiety; distraction of attention; child
MeSH Terms: conditions — Dyspnea; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two groups with traditional therapy control group.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- virtual reality (Experimental): Pre-Procedure: Information about the study will be given. Children with a pain score of '0' will be included in the groups. Verbal and written consent will be obtained from those who voluntarily agree to participate in the study. Video recording will be started with a mobile phone. Physiological parameters and anxiety level of the children will be measured and recorded 1 minute before the treatment. HFNC oxygen therapy will be started with video demonstration accompanied by virtual reality glasses. Physiological parameters and anxiety level will be recorded 10 minutes after HFNC oxygen treatment. Video recording will be terminated. Since the parameters in the scales should be evaluated by 2 nurses independent of the study during the study, only the behaviours of the child during the procedure should be video recorded by means of a mobile phone. For participants and parents who want to participate in the study but do not approve the video recording, the parameters will be evaluated ins
  Interventions: Device: Virtual reality goggles during HFNC
- routine procedure (Active Comparator): Information about the study will be given. Children with a pain score of '0' will be included in the groups. Verbal and written consent will be obtained from those who voluntarily agree to participate in the study. Video recording will be started with a mobile phone. Physiological parameters and anxiety level of children will be measured and recorded 1 minute before the treatment. HFNC oxygen therapy will be started with routine ward practice. Physiological parameters and anxiety level will be recorded 10 minutes after HFNC oxygen treatment. Video recording will be terminated. Since the parameters in the scales should be evaluated by 2 nurses independent of the study during the research, only the behaviours of the child during the procedure should be video-recorded by means of a mobile phone. For participants and parents who want to participate in the study but do not approve the video recording, the parameters will be evaluated instantly by a researcher independent from the study.
  Interventions: Device: HFNC oxygen therapy with routine service application

INTERVENTIONS:
Device: Virtual reality goggles during HFNC — HFNC oxygen therapy will be started with video demonstration accompanied by virtual reality glasses. Physiological parameters and anxiety level will be recorded 10 minutes after HFNC oxygen treatment. Video recording will be terminated. Since the parameters in the scales should be evaluated by 2 nurses independent of the study during the study, only the behaviours of the child during the procedure should be video recorded by a mobile phone. For the participants and parents who want to participate in the study but do not approve the video recording, the parameters will be evaluated instantly by a researcher independent from the study. The study will continue until the 30-person intervention group is completed.
  Arms: virtual reality
Device: HFNC oxygen therapy with routine service application — HFNC oxygen therapy will be started with routine ward practice. Physiological parameters and anxiety level will be recorded 10 minutes after HFNC oxygen treatment. Video recording will be terminated. Since the parameters in the scales should be evaluated by 2 nurses independent of the study during the research, only the behaviours of the child during the procedure should be video-recorded by means of a mobile phone. For participants and parents who want to participate in the study but do not approve the video recording, the parameters will be evaluated instantly by a researcher independent from the study
  Arms: routine procedure

SUMMARY:
Determination of the effect of virtual reality goggles used during high-flow oxygen therapy on child anxiety in children

DETAILED DESCRIPTION:
Respiratory system diseases are frequently seen in childhood and hospitalised constitute a significant portion of the applications. Children continue their treatment in paediatric clinics or intensive care units according to their clinical conditions. In paediatric intensive care units, patients need respiratory support at various rates and respiratory support therapies are among the most commonly used treatment methods in paediatric intensive care clinics. Oxygen given to the appropriate patient under appropriate conditions treatment accelerates the healing process of the disease and prevents the progression of the current situation in a bad course and reduces mortality and morbidity. Oxygen therapy in hospitalised children invasive or non-invasive methods. Invasive method is the treatment method in which endotracheal intubation and mechanical ventilator are used. Noninvasive oxygen therapies are basically analysed in two groups as low-flow and high-flow applications. Low flow oxygen therapy is applied with nasal cannula, hood and tent system, simple face mask, reservoir mask and diffuser mask. High-flow oxygen systems include venturi mask, continuous positive airway pressure (cpap) therapy, bi-level positive airway pressure (bipap) therapy and high-flow nasal cannula oxygen therapy (HFNC). HFNC therapy is a non-invasive form of respiratory support that allows the delivery of high flow (30-60 L/min) of humidified and heated air (31 to 37°C) at a certain oxygen concentration (21-100%) through a nasal cannula, which can be used in the treatment of acute and chronic diseases with values appropriate to the patient's age/body weight and needs. Compared to normal nasal cannula and face mask, HFNC provides a higher level of respiratory support.

can happen. Children experience discomfort and anxiety due to the pressure created by the flow rate and the sound made by the device, and discomfort from the nasal cannula causes resistance to treatment. Nurses are responsible for implementing HFNC, observing the effectiveness of the treatment, monitoring children during HFNC and maintaining their daily life activities, and in this process, they benefit from evidence-based nursing practices. Medical procedures encountered during hospitalisation are the main source of fear for children. They may experience anger, helplessness and anxiety due to reasons such as unfamiliar environment, change in the routine of the child, different sound, light, tools and equipment, unfamiliar people, painful painful procedures, being away from family and friends, loss of control, activity limitation, communication difficulties, presence of other children crying. The use of technology in preparation for or during medical procedures is an effective method in providing anxiety and comfort. At the same time, respiratory distress experienced by children causes anxiety, dyspnoea and increased respiratory rate. In addition to the provision of effective respiratory support, it is important to improve children's experience of the hospital process and In order to support long-term physical and psychosocial health, it is necessary to utilise distraction methods for anxiety management. Nurses is independently involved in the management of oxygen therapy to prevent and protect patients from the adverse effects of hypoxaemia. Distraction methods, atraumatic care It is one of the non-pharmacological methods among the approaches and is used to control pain, stress and anxiety. There are many methods used to divert attention.

Some of them are; watching cartoons, hypnotherapy, playing with toys, using virtual reality, music therapy, play therapy, using kaleidoscope and using distraction cards. This study was planned to determine the effect of virtual reality used during high flow nasal cannula oxygen therapy on physiological parameters and anxiety levels in children aged 6-12 years.

ELIGIBILITY:
Inclusion Criteria:

* The child is between 6-12 years old
* The child is receiving high flow nasal cannula oxygen therapy in the paediatric intensive care unit
* The child has no visual and hearing problems
* No pain according to the Wong-Baker pain scale
* No genetic, congenital, chronic or metabolic disease
* Being conscious and able to communicate verbally
* Written and verbal acceptance of the child and his/her parents to participate in the study after the information.

Exclusion Criteria:

* The child is in pain.
* The child is taking a sedative medication
* The child has a fever above 37°C
* The child presented with a severe asthma attack
* The child's saturation value was below 92% at the time of admission

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Children's Emotional Manifestation Scale-CEMS | 1 minute before the start of the procedure and 1 minute after 10 minutes of VR viewing
  It was developed in 2003 by William Li and Lopez to assess the level of anxiety in children aged 7-12 years. The Turkish validity and reliability of the scale was carried out by Yanık et al. in 2019 with the approval and opinion of William Li and Lopez on the appropriateness of evaluating anxiety in children aged 3-6 years. The scale has 5 different categories and 25 items and is used to assess the anxiety level of children aged 3-12 years during medical interventions. In the facial expression category, the facial expressions of the child are evaluated by the researcher. In the vocalisation category, tear status is evaluated. In the movement category, the child's body language is evaluated. In the interaction category, the child's verbal/non-verbal communication status is evaluated. In the cooperation category, the child's active / passive participation is evaluated. Each category is between 1-5 points and a total score between 5-25 points is obtained. Cronbach's Alpha value is 0.969.

SECONDARY OUTCOMES:
Wong and Baker Faces Pain Scale | immediately before starting the process
  This scale was developed by Donna Wong and Connie Morain Baker in 1981 and revised in 1983 and is a tool used to assess the level of pain in children aged 3-18 years who can communicate. In this scale, face shapes are used for children to express their pain level. Each face shape has a numerical equivalent. In the scale, the lowest pain level is evaluated as '0' and the highest pain level is evaluated as '10'. As the level of pain increases, the intensity of the pain increases numerically and is expressed by facial expression.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba KARAKUŞ TÜRKER, Study Director — Üsküdar University Faculty of Health Sciences
Locations (1):
- Şehit Prof. Dr. İlhan Varank Sancaktepe Training and Research Hospital, Istanbul, Sancaktepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I'll share it if necessary, I'm not thinking about it now.